CLINICAL TRIAL: NCT05992194
Title: Exploratory Study Analyzing the Repeatability of Neurovisual Tasks for the Construction of a New Concussion Monitoring Tool
Brief Title: Repeatability Assessment of Neurovisual Tasks for the Construction of a New Concussion Monitoring Tool (SPORTICARE)
Acronym: SPORTiCARE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SBN_2023_2
Record Dates: First submitted 2023-08-04; First posted 2023-08-15 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: multimodal oculomotor measurements — * Visual assessment to ensure that the subject meets the inclusion and non-inclusion criteria, including anamnesis and the following visual tests: Lang stereotest, H-test ocular motility, convergence, masking and accommodative rock.
  * Evaluation by experimenter A (60 min)
    * Neuro-ophthalmological tests on screen
    * Neuro-ophthalmological tests in VR headset
  * Evaluation by experimenter B (60 min)
    * Neuro-ophthalmological tests on screen
    * Neuro-ophthalmological tests in VR helmet The sequence of experimenters A-B or B-A will be randomized.

SUMMARY:
Traumatic brain injury (TBI) is a condition that occurs when a mechanical blow to the head causes damage to the brain. The diagnosis of this pathology requires the evaluation of several dimensions, including clinical symptoms, physical signs, cognitive disorders, behavioral and sleep disturbances and state of consciousness. This multidimensional approach provides a comprehensive and accurate assessment of head injury and its severity.

The Berlin Consensus of the International Conference on Concussion in Contact Risk Sports held in Berlin in 2016 (McCrory et al., 2017) emphasized that the management of a CTE must be multimodal and multidisciplinary.

This expert consensus converged on a tool that is now the most widely used in protocols studying concussion in sports at risk of BTI. This tool, the SCAT 5 (Sports Concussion Assessment Tool), combines symptom assessment, cognitive examination, neurological examination (oculomotricity, balance) and immediate and delayed memory.

However, it requires the intervention of a medical expert to assess the clinical signs of the concussed athlete. Hänninen et al (2021) showed that test-retest reproducibility was very good for the clinical symptomatology subscore, but poor or average for the subscores summarizing cognitive tests and balance assessment.

Clinicians now need to be able to better assess the severity of damage following head injury, and to monitor the patient's progress. This will improve the management of concussed athletes right up to their eventual return to sporting activity.

The ultimate aim of our project is to develop and optimize an easily exportable multimodal concussion assessment tool, based on the use of a virtual reality headset, which will enable us to objectively characterize the state and evolution of a subject after a TCE. This will enable the assessment of neuro-visual functions and compensations in the concussed patient, revealing a higher attentional cost characterized by instability of orthostatic control, higher blink frequency and larger pupil size.

The multimodal tool will be built from the results of various tests:

* Standardized oculomotor tasks(pro-saccades, anti-saccades, smooth pursuit, memory guided saccades, self paced saccades)
* Orthostatic balance control to assess postural compensations and estimate attentional cost during oculomotor tasks.
* Pupil dynamics using the Pupil Cycle Time (PCT) test. The aim of this exploratory study is to determine the repeatability of measurements provided by the SPORTiCARE virtual reality headset during different tasks.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity of 10/10,
* Express consent to participate in the study,
* Affiliated (or beneficiary) of a social insurance scheme.

Exclusion Criteria:

* History of Cranioencephalic Trauma,
* Protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure (guardianship or curatorship).
* Subjects suffering from a degenerative disease or any other illness which could interfere with the evaluations planned during this study (migraine, balance disorders, vertigo).
* Subjects with ophthalmological pathologies affecting visual functions (oculomotor dysfunction, diplopia, strabismus).
* Known history of convergence and/or accommodation insufficiency.
* Subject declaring to the investigator in charge of anamnesis, consumption of psychoactive and psychotropic drugs, medications (anti-anxiety, antidepressant, anticonvulsant, opiate, analgesic, anti-hypertensive) or level 3 medications, which may have effects on vision.
* Unavailability of participant for evaluation sessions.
* Inability to comply with study task instructions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group of 25 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Assessment of repeatability when performing pro-saccades | Day 0
  Latency (ms)
Assessment of repeatability when performing anti-saccades | Day 0
  Latency (ms)
Assessment of repeatability when performing memory tricks | Day 0
  Positional error (degrees)
Assessment of repeatability of the number of saccades when performing self-paced saccades | Day 0
  number of saccades (n) performed between the two targets in the allotted time (15 seconds)
Assessment of repeatability of pupil cycle time when performing self-paced saccades | Day 0
  Pupil Cycle Time (PCT): average frequency of pupillary oscillation (Hz)
Assessment of repeatability when performing pro-saccades | Between Day 7 and Day 21
  Latency (ms)
Assessment of repeatability when performing anti-saccades | Between Day 7 and Day 21
  Latency (ms)
Assessment of repeatability when performing memory tricks | Between Day 7 and Day 21
  Positional error (degrees)
Assessment of repeatability of the number of saccades when performing self-paced saccades | Between Day 7 and Day 21
  number of saccades (n) performed between the two targets in the allotted time (15 seconds)
Assessment of repeatability of pupil cycle time when performing self-paced saccades | Between Day 7 and Day 21
  Pupil Cycle Time (PCT): average frequency of pupillary oscillation (Hz)

CONTACTS AND LOCATIONS:
Locations (1):
- Streetlab - Institut de la Vision, Paris, France

IPD SHARING:
Plan to Share IPD: No